CLINICAL TRIAL: NCT01191177
Title: An Initial Trial of Enteral Fish Oil Supplementation in the Treatment of Parenteral Nutrition-associated Liver Disease in Patients With Short Bowel Syndrome
Brief Title: Investigational Study of Oral Fish Oil in Treating Parenteral Nutrition Associated Liver Disease
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: no subjects recruited
Sponsor: Boston Children's Hospital (Other)
Collaborators: Harvard University (Other); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Tom Jaksic, W. Hardy Hendren Professor of Surgery, Harvard Medical School, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-02-0066
Record Dates: First submitted 2010-08-27; First posted 2010-08-30 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Liver Disease; Short Bowel Syndrome
Keywords: oral fish oil; Lovaza; Omega-3-acid supplementation
MeSH Terms: conditions — Liver Diseases; Short Bowel Syndrome | interventions — Omacor; Fish Oils; Corn Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lovaza group (Experimental): Patients randomized to this group will receive Lovaza 1gram per kilogram of body weight, not exceeding 4grams a day
  Interventions: Drug: Lovaza (omega-3-acid ethyl ester)
- Placebo group (Placebo Comparator): Patients randomized to this group will receive corn oil supplement 1gram per kilogram of body weight, not exceeding 4grams per day
  Interventions: Dietary Supplement: Corn oil

INTERVENTIONS:
Drug: Lovaza (omega-3-acid ethyl ester) — supplied as 1gram transparent soft-gelatin capsules filled with yellow oil, dosage is 1gram per kilogram of body weight per day, not exceeding 4grams per day until normalization of liver function test
  Other Names: fish oil
  Arms: Lovaza group
Dietary Supplement: Corn oil — 1 gram per kilogram body weight per day, not exceeding 4 grams
  Arms: Placebo group

SUMMARY:
The purpose of this study is to investigate the usefulness of oral fish oil(Lovaza)in normalizing liver function in patients who have parenteral nutrition associated liver disease. The investigators believe that patients who take oral fish oil will normalize liver function faster than those who do not

DETAILED DESCRIPTION:
This is designed as a randomized placebo controlled trial of oral fish oil (Lovaza) in normalizing parenteral nutrition associated liver disease.

ELIGIBILITY:
Inclusion Criteria:

* History of parenteral nutrition(PN)administration >4weeks
* PN associated liver disease from intestinal failure
* ability to take full enteral feed
* body weight equal or greater than 3kg
* elevated ALT level twice of that normal(ALT>84)at the time PN is weaned off

Exclusion Criteria:

* Hemodynamic instability
* renal failure
* suspected congenital obstruction of the hepatobiliary system
* diagnosis hepatitis A, B, or C
* diagnosis of alpha 1-antitrypsin deficiency
* diagnosis of cytomegalovirus infection
* diagnosis of HIV
* children in care

Ages: 30 Days to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Normalization of ALT
  The primary aim is to examine the efficacy of Lovaza, when compared to placebo, on normalizing liver function, as measured primarily by amino alanine transferase (ALT). The investigators believe that patients in the Lovaza group will normalize ALT faster than in the placebo group.

SECONDARY OUTCOMES:
Normalization other liver function tests and inflammatory status
  The investigators believe that Lovaza will result in faster reduction of the serum levels of the following markers: total bilirubin, aspartate amino transferase (AST), alkaline phosphatase, gamma glutamyl transpeptidase (GGTP) & C-reactive protein (CRP).

CONTACTS AND LOCATIONS:
Overall Officials: Tom Jaksic, MD, PhD, Principal Investigator — Children's Hopsital Boston
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No